CLINICAL TRIAL: NCT05883540
Title: Lysergic Acid Diethylamide (LSD) in Palliative Care: a Randomised, Double-blind, Active-placebo Controlled Phase II Study (LPC-Study)
Brief Title: Lysergic Acid Diethylamide (LSD) in Palliative Care
Acronym: LPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital, Zürich (Other); Spital Uster AG, Uster, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BASEC 2022-01818
Record Dates: First submitted 2023-05-08; First posted 2023-06-01 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Palliative Care; Pain; Anxiety; Depression; Demoralization; Psychological Distress; Quality of Life; Caregiver Burden; Fear of Death; Existential Distress
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression; Caregiver Burden; Necrophobia | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment arm (Experimental): Subjects in the treatment arm will receive 100 μg LSD (first session) and 100 or 200 μg LSD (second session) per os.
  Interventions: Drug: Lysergic Acid Diethylamide Tartrate
- control arm (Active Comparator): Subjects in the control arm will receive 25 μg LSD (first session) and 25 μg LSD (second session) per os.
  Interventions: Drug: Lysergic Acid Diethylamide Tartrate

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide Tartrate — 25 μg p.o.
  Other Names: LSD
  Arms: control arm
Drug: Lysergic Acid Diethylamide Tartrate — 100 or 200 μg p.o.
  Other Names: LSD
  Arms: treatment arm

SUMMARY:
Background: Terminally ill patients often experience significant psychosocial distress having depressed mood, death anxiety, pain, and an overall poor quality of life. Recent evidence from pilot studies suggests that serotonergic hallucinogens including lysergic acid diethylamide (LSD) and psilocybin produce significant and sustained reductions of depressive symptoms and anxiety, along with increases in quality of life, and life meaning in patients suffering from life-threatening diseases. Additionally, serotonergic hallucinogens may produce antinociceptive effects.

Objective and Design: The study aims to evaluate effects of LSD on psychosocial distress in 60 patients suffering from an end-stage fatal disease with a life expectancy ≥12wks and ≤2yrs in an active placebo-controlled double-blind parallel study. Patients will be allocated in a 2:1 ratio to one of the two intervention arms receiving either two moderate to high doses of LSD (100 µg and 100 µg or 100 µg and 200 µg) as intervention and two low doses of LSD (25 µg and 25 µg) as active-placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years.
* End-stage fatal disease of any cause with a life expectancy ≥ 12 weeks and ≤ 2 years
* Sufficient understanding of the study procedures and risks associated with the study.
* Participants must be willing to adhere to the study procedures and sign the consent form.
* Participants must be willing not to drive a traffic vehicle or to operate machines within 24 h after LSD administration.
* Participants must complete an actual "Emergency Medical Directive"

Exclusion Criteria:

* Life expectancy < 12 weeks
* Known hypersensitivity to LSD
* Requiring ongoing concomitant therapy with a psychoactive prescription drug which might interfere with the study drug, and unable or unwilling to comply with the washout period.
* Current use of a potent drug CYP2D6 inhibitor
* Women who are pregnant or nursing or intend to become pregnant during the course of the study.
* Somatic disorders including CNS involvement of cancer, untreated epilepsy with a history of grand-mal seizures, history of delirium, end-stage heart failure (NYHA IV), untreated hypertension or insufficiently treated hypertension, angina pectoris, severe liver disease or severely impaired renal function, or other that in the judgement of the investigators pose too great potential for side effects.
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant.
* Participation in another study with an investigational drug within the 30 days preceding and during the present study
* concomitant diagnosis of past or present psychotic disorder, first-degree relative with psychotic disorders
* concomitant diagnosis of past or present bipolar disorder
* current delirium
* substance use disorder (within the last 2 months, except nicotine, opioids used for analgesia, and benzodiazepine treatment for anxiety).
* Weight < 45 kg
* Suicidal ideation with active intent or plan to act on suicidal thoughts as assessed by the treating investigator.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Changes in state anxiety assessed by questionnaire (state anxiety inventory, STAI-S) compared with active placebo | baseline, 2 weeks after second intervention
  State anxiety inventory (STAI-S) scores, 20 items

SECONDARY OUTCOMES:
Changes in state anxiety assessed by questionnaire (state anxiety inventory, STAI-S) compared with active placebo | baseline, 2 days after each intervention, 4 weeks, 6 weeks, and 9 weeks after second intervention
  State anxiety inventory (STAI-S) scores, 20 items
Changes in pain levels assessed by questionnaire compared with active placebo | baseline, 2 days after each intervention and 2 weeks after second intervention; 4 weeks, 6 weeks, and 9 weeks after second intervention
  numeric rating scale (NRS) scores ranging from 0 (no pain) to 10 (maximum imaginable pain)
Changes in opioid use (dosages of opioids unified according to equivalent dosages of oral morphine) compared with active placebo | concomitant medication will be assessed several times over whole study duration up to 9 weeks after second intervention
Changes in spiritual well-being assessed by questionnaires (Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being; The 12-item Spiritual Well-Being Scale (FACIT-Sp-12)) compared with active placebo | baseline, 2 days after each intervention and 2 weeks after second intervention; 4 weeks, 6 weeks, and 9 weeks after second intervention
  Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being; The 12-item Spiritual Well-Being Scale (FACIT-Sp-12) scores
Changes in demoralization assessed by questionnaires (Demoralization Scale II (DS-II)) compared with active placebo | baseline, 2 days after each intervention and 2 weeks after second intervention; 4 weeks, 6 weeks, and 9 weeks after second intervention
  Demoralization Scale II (DS-II) scores
Changes in quality of life assessed with a single-item question compared with active placebo | baseline, 2 days after each intervention and 2 weeks after second intervention; 4 weeks, 6 weeks, and 9 weeks after second intervention
  single-item question "how satisfied are you currently with your physical and emotional well-being" rated on a 7-point scale (1 dissatisfied, 7 satisfied)
Changes in anxiety, pain levels, quality of life, demoralization, and spiritual well-being shortly after first intervention compared with scores shortly after second intervention | post drug visit 1-3 compared with post drug visit 4-6
  State anxiety inventory (STAI-S), NRS, QoL single-item, Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being; The 12-item Spiritual Well-Being Scale (FACIT-Sp-12), and Demoralization Scale II (DS-II) scores
Changes in patient's depression, isolation, anxiety, fear and denial of imminence of death, and pre-occupation with pain using investigator-ratings compared with active placebo | baseline, one day before second intervention and 2 and 9 weeks after second intervention
  Emotional Condition Rating Scale (ECRS) scores, Hamilton depression (GRID-HAM-D17) and Hamilton anxiety rating scale (HAM-A) scores
Changes in patient's behaviour and attitudes rated by community observers compared with active placebo | baseline, before second intervention and 2 weeks and 9 weeks after second intervention
  community observer rating: rating of the participant's behaviour and attitudes on 11 items by a contact person
Changes in caregiver burden assessed by questionnaire compared with active placebo | baseline, before second intervention and 2 weeks and 9 weeks after second intervention
  Zarit Burden Inventory (ZBI) scores completed by caregiver, total score
Associations between acute LSD effects assessed with questionnaires and long-lasting therapeutic effects assessed with questionnaires | 2,4,6, and 9 weeks after second intervention
  acute effects will be assessed using the Mystical experience Questionnaire (MEQ30) and visual analogue scales (VASs)
Changes in burden of suffering assessed with the Pictorial Representation of Illness and Self-Measure (PRISM) compared with active placebo | baseline, 2 days after each intervention, 2 weeks and 9 weeks after the second intervention
Qualitative description of subjective changes after intervention assessed with semistructured interviews | baseline, 2 days after each intervention, 2 weeks and 9 weeks after second intervention
Expectancy as a mediator for treatment effects assessed with questionnaire | baseline
  modified version of the Credibility / Expectancy Questionnaire (CEQ)
Assessment of adverse events (AE) | during the whole study duration up to 9 weeks after second intervention
  grading according to Common Terminology Criteria for Adverse Events CTCAE Version 5.0, safety measures
Physical and general discomfort during drug sessions using standardized questions (adapted list of complaints) | before and 12 hours after drug administration
  adapted list of complaints (LC), safety measures
Changes in vital signs during drug sessions | before and up to 12 hours after drug administration
  monitoring blood pressure and heart rate with an automatic oscillometric device, safety measure
Changes in vital signs during drug sessions | before and up to 12 hours after drug administration
  monitoring body temperature using an ear thermometer, safety measure

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Schmid, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (3):
- Switzerland (3):
  - Spital Uster AG, Uster, Canton of Zurich
  - University Hospital Basel, Basel
  - University Hospital Zurich, Clinic for Radio-Oncology, Competence Centre Palliative Care, Zurich

REFERENCES:
- [Derived] Schipper S, Nigam K, Schmid Y, Piechotta V, Ljuslin M, Beaussant Y, Schwarzer G, Boehlke C. Psychedelic-assisted therapy for treating anxiety, depression, and existential distress in people with life-threatening diseases. Cochrane Database Syst Rev. 2024 Sep 12;9(9):CD015383. doi: 10.1002/14651858.CD015383.pub2. PMID 39260823